CLINICAL TRIAL: NCT00053976
Title: Treatment of Acute Graft vs. Host Disease With Steroids Plus Daclizumab (Zenapax) or Placebo
Brief Title: Methylprednisolone With or Without Daclizumab in Treating Patients With Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, VIncent T. Ho, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99-279; P30CA016056 (NIH); P30CA006516 (NIH); RPCI-DS-0218; ROCHE-RPCI-DS-0218
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Daclizumab; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daclizumab (Experimental): Patients are randomized to 1 of 2 treatment arms.
  Arm I:
  * Patients receive methylprednisolone or equivalent corticosteroid IV or orally
  * Daclizumab IV on days 0, 3, 7, 14, and then weekly as indicated until day 100.
  Arm II: Patients receive methylprednisolone or equivalent corticosteroid as in arm I and placebo.
  Patients are followed at 1 year and then annually thereafter.
  Interventions: Biological: Daclizumab; Drug: methylprednisolone
- Placebo (Placebo Comparator): Patients are randomized to 1 of 2 treatment arms.
  * Patients receive methylprednisolone or equivalent corticosteroid as in Daclizumab arm
  * Placebo IV on days 0, 3, 7, 14, and then weekly as indicated until day 100.
  Interventions: Drug: methylprednisolone; Drug: Placebo

INTERVENTIONS:
Biological: Daclizumab
  Other Names: Zenapax
  Arms: Daclizumab
Drug: methylprednisolone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of IL2 receptor antibody (also known as Daclizumab or Zenapax) and corticosteroids alone for control of GVHD. Treatment with corticosteroids is standard care for GVHD. This research is being done because the investigators do not know whether addition of this new medication to standard corticosteroid therapy improves response rates. Since Zenapax binds to a type of cell which is thought to cause GVHD and possibly inactivates them, investigators have reason to believe that addition of Zenapax night result in better control of GVHD This study will determine whether the addition of another medication, Zenapax, will be more effective than steroids alone in suppressing GVHD and improving symptoms of GVHD.

Daclizumab (Zenapax) is approved by the Food and Drug Administration (FDA) for use in patient with kidney transplant to help prevent graft rejection. This medication has been used in bone marrow transplant patients to treat GVHD.

DETAILED DESCRIPTION:
GVHD occurs when the donor's immune system recognizes a patient's body as foreign and reacts against it. GVHD may result in skin rashes and blistering, liver inflammation and gastrointestinal problems including nausea, vomiting, diarrhea and bleeding. Mild GVHD may be treated with topical medications applied to the skin. More severe GVHD requires medications given intravenously (by vein) or taken by mouth. Steroids are usually given first to treat GVHD but only 40% of people respond to this alone.

OBJECTIVES:

* Compare response to treatment in patients with acute graft-versus-host disease (GVHD) treated with methylprednisolone with or without daclizumab.
* Compare differences in total methylprednisolone dose and complications in patients treated with these regimens.
* Compare mortality, days of antibiotics and antifungal therapy, and required hospital days within the first 100 days for patients treated with these regimens.
* Compare overall survival and incidence of chronic GVHD at 1 year in patients treated with these regimens.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to prior graft-versus-host disease (GVHD) prophylaxis (immunosuppressive therapy vs T-cell depletion), GVHD organ manifestation (skin only vs other), donor type (6/6 matched sibling vs other), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive methylprednisolone or equivalent corticosteroid IV or orally and daclizumab IV over 15 minutes on days 0, 3, 7, 14, and then weekly as indicated until day 100.
* Arm II: Patients receive methylprednisolone or equivalent corticosteroid as in arm I and placebo.

Patients are followed at 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria

* Allogeneic Transplantation
* Acute GVHD requiring therapy (skin stage 2 or overall grade II-IV)
* Signed, informed consent

Exclusion Criteria

* Mental or emotional contraindications as determined by patient's physician
* Steroids given prophylactically or therapeutically at a dose > 1 mg/kg/d methylprednisolone (including prevention of acute GVHD or treatment for diffuse alveolar hemorrhage and severe obstructive mucositis within 7 days prior to starting acute GVHD therapy. Steroids administered as amphotericin premedication are allowed if below 1 mg/kg/day.
* Acute GVHD diagnosed solely by virtue of upper GI GVHD
* Hypersensitivity to Daclizumab or prior therapy with Daclizumab
* GVHD from donor lymphocyte infusion
* Other investigational therapeutics within 30 days of enrollment
* Pregnancy or of fertile, failure to agree to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-01; Primary Completion 2003-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Rate of decrease of acute GVHD grade | Day 42

SECONDARY OUTCOMES:
100 Day Mortality | 100 Day
Complete Response of GVHD | 100 Days
Total Days of Antibiotic or Antifungal | 100 Days
Number of Hospitalized Days | 100 Days
Total Steroid Dose | 100 Days
Number of Participants with Steroid related Complication | 1 Year
Overall Survival | 100 Days
Relapse Rate | 1 Years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J. Lee, MD, Study Chair — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No